CLINICAL TRIAL: NCT03962335
Title: ModulAtion of Gut Microbiota Through Nutritional Interventions in Behcet's Syndrome pAtients: the MAMBA Study
Brief Title: Gut Microbiota and Behcet's Syndrome: a Dietary Intervention Trial (MAMBA Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Ospedaliero-Universitaria Careggi (Other)
Responsible Party: Principal Investigator, Francesco Sofi, Associate Professor of Clinical Nutrition, Azienda Ospedaliero-Universitaria Careggi
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MAMBA
Record Dates: First submitted 2019-05-14; First posted 2019-05-24 (Actual); Last update posted 2024-02-02 (Actual); Status verified 2024-02

CONDITIONS: Behcet Syndrome
Keywords: Gut microbiota; Mediterranean diet; Vegetarian diet; Short chain fatty acids
MeSH Terms: conditions — Behcet Syndrome | interventions — Diet, Vegetarian; Diet, Mediterranean; Butyrates

STUDY DESIGN:
Intervention Model Description: Randomized crossover open dietary intervention study with 3 arms of intervention
Masking Description: In this trial blinding of participants and investigators will not be possible because of obvious differences between the intervention diets
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VD group (Experimental): Group that starts with Vegetarian diet (VD)
  Interventions: Behavioral: Vegetarian diet; Behavioral: Mediterranean diet with butyrate; Behavioral: Mediterranean diet
- MD+Bt group (Experimental): Group that starts with Mediterranean diet with oral supplementation with butyrate (MD+Bt)
  Interventions: Behavioral: Vegetarian diet; Behavioral: Mediterranean diet with butyrate; Behavioral: Mediterranean diet
- MD group (Active Comparator): Group that starts with Mediterranean diet (MD)
  Interventions: Behavioral: Vegetarian diet; Behavioral: Mediterranean diet with butyrate; Behavioral: Mediterranean diet

INTERVENTIONS:
Behavioral: Vegetarian diet — 7-days dietary profile with a Vegetarian diet (VD), containing inulin and resistant starch-rich foods and including no meat and fish, but containing eggs and dairy, for 3 months
  Other Names: VD
Behavioral: Mediterranean diet with butyrate — 7-days dietary profile with Mediterranean diet with oral supplementation with butyrate (MD+Bt), 2 g/day, for 3 months
  Other Names: MD+Bt
Behavioral: Mediterranean diet — 7-days dietary profile with Mediterranean diet (MD), including 2 portions per week of fish and 3 portions per week of fresh and processed meat (2 of which fresh or processed red meat), for 3 months
  Other Names: MD

SUMMARY:
Behçet's syndrome (BS) is an idiopathic, chronic, multi-systemic inflammatory disorder characterized by ocular disease, skin lesions, vascular, neurological and gastrointestinal involvement. A recent study showed a peculiar dysbiosis of gut microbiota (GM) in BS patients, with specific changes in the profiles of short-chain fatty acids, especially butyrate. Over the last few years, a growing interest on the role of GM in metabolic disturbances has been manifested. Diet is one of the major factors driving the GM composition and functionality. In this context, the influence of diets generally recognized healthy on GM has been explored, but consistent data on autoimmune and inflammatory diseases are not available. The aim of this intervention study is to investigate whether a lacto-ovo-vegetarian diet enriched in substrates with potential for butyrate production or a Mediterranean diet supplemented with oral butyrate could be beneficial for GM and metabolic risk profile in BS.

DETAILED DESCRIPTION:
Background / State of Art:

Behçet's syndrome (BS) is a systemic inflammatory disorder characterized by a wide range of potential clinical manifestations with no gold-standard therapy. Although BS is usually not a life-threatening condition, mortality can be associated with vascular-thrombotic and neurological affections.

A recent study by our group, for the first time, provided evidence of a peculiar gut microbiota (GM) dysbiosis in BS patients, with reduced biodiversity, and decrease in short-chain fatty acid (SCFA)-producers and butyrate production. In light of this, controlled dietary interventions specifically designed to favor the increase of butyrate-producing members of the GM may support the recovery of a healthy GM ecosystem. Lacto-ovo-vegetarian diet is characterized by abstention from consuming meat and meat products, poultry, seafood and flesh from any other animal and by a large amount of plant- derived foods. This dietary pattern has been largely demonstrated to be beneficial for both patients with an established disease and for subjects with traditional risk factors for chronic diseases. Indeed, dietary patterns rich in plant-based food have been found to promote a more favorable GM profile, according to the high amount of dietary fiber and fermentable substrate, which are sources of metabolic fuel for GM fermentation that, in turn, result in end products - mainly SCFA - that are key microbial metabolites with a multifactorial role on the host health.

Hypothesis and Specific aims:

Although the pathogenesis of BS is currently unknown, it has been recently classified at the crossroad between autoimmune and autoinflammatory syndromes. GM has been found to deeply influence our metabolic and immunological health, and specific perturbed GM configurations have been indicating a fascinating link between intestinal microbes and health status. A recent study from our group showed that a peculiar dysbiosis of the GM ecosystem is present also in patients with BS, corresponding to specific changes in the profiles of SCFA production. In particular, the GM ecosystem in BS showed a low biodiversity, in line with several other chronic disorders. Moreover, a significant depletion of well- known butyrate producers, Roseburia and Subdoligranulum, and a corresponding decrease of butyrate production in BS patients was demonstrated. Butyrate - which is the preferred fuel for colonocytes - is able to induce T regulatory cell differentiation via several mechanisms, so the butyrate impairment in BS patients could favor a reduced T regulatory cell- mediated control, thus promoting a powerful immuno-pathological T cell responses.

In this context, over the last years, growing evidence suggested that high-fiber dietary patterns are able to promote a more favorable GM profile, and are key mediators of microbial diversity. In particular, it has recently been demonstrated that high adherence to a lacto-ovo-vegetarian diet - including high intake of non-refined cereals, fruit, vegetables and legumes - is associated with a beneficial GM profile, with enrichment in fiber-degrading bacteria and increase of fecal SCFA. In a similar way, other dietary patterns have been shown to modulate GM dysbiosis, by supporting the recovery of a balanced microbial community of health-promoting SCFA-producing members with the decrease of pro-inflammatory groups. Furthermore, current evidence indicates that the consumption of certain fibers - such as inulin and resistant starch - leads to specific GM rearrangements with the production of more butyrate than others in humans.

All these findings let hypothesize that the adherence to a controlled dietary profile such as lacto-ovo-vegetarian diet, possibly enriched in substrates with potential for butyrate production may select butyrate-producing bacteria - especially Roseburia spp. (Clostridium cluster XIVa) and Faecalibacterium prausnitzii (Clostridium cluster IV)- so reversing the pro- inflammatory dysbiosis observed in BS.

Preliminary Data:

A recent study by our group showed that a peculiar dysbiosis of the GM ecosystem is present in patients with BS, corresponding to specific changes in the profiles of SCFA production. By strengthening this dysbiotic GM structure, a significant decrease of fecal butyrate production was found in BS patients. More recently, a high percentage of Th1/Th17 cells at gut mucosal level in BS patients was observed, thus suggesting a reduced T regulatory activity, probably mediated by reduced levels of butyrate (unpublished data).

Specific Aim 1: To conduct a dietary intervention randomized controlled trial in order to investigate whether a lacto-ovo-vegetarian diet enriched in substrates with potential for butyrate production or a Mediterranean diet supplemented with 2 g/day of butyrate could be beneficial for GM and for the amelioration of the clinical manifestations and disease severity of patients with BS.

Specific Aim 2: To evaluate the effects of these interventions on: inflammatory parameters, circulating biomarkers of disease, endogenous butyrate production, and oxidative stress markers.

Specific Aim 3: To validate and extend our preliminary results on GM ecosystem dysbiosis in BS patients

ELIGIBILITY:
Inclusion Criteria:

* Behcet syndrome
* Age 18-65 years
* Willing to give informed consent
* Willing to participate in a study where one of the proposed dietary profile is a vegetarian pattern

Exclusion Criteria:

* Pregnancy or lactation
* Concomitant presence of serious illness or unstable condition (autoimmune diseases; chronic viral infections; malignancies, recent myocardial infarction, chronic liver disease, inflammatory bowel diseases)
* Current or recent (past 6 months) participation in weight loss treatment program or use of weight loss medication
* Adoption of a vegetarian diet for the past 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Disease severity of Behcet syndrome assessed by Behçet Disease Current Activity Form | 1 year
  The disease activity will be assessed by the use of the validated Behçet Disease Current Activity Form (BCDAF), at the baseline and after the dietary intervention. The BCDAF will assess the presence of oral and genital ulceration, skin, joint and gastrointestinal involvement, presence of fatigue and headache with a 5-point scale according to the duration of symptoms, with 0 meaning no symptoms and 4 meaning symptoms for 4 weeks. The presence of eyes, large vessels or central nervous system (CNS) involvement are document with "yes/no" answers. In addition, patients will be asked to rate on a 7-point scale how active they felt. Similarly, the clinicians will complete a 7-rating scale to assess their opinion of overall activity of the disease, with lower scores representing better outcomes.
Behcet disease's improvement of symptoms assessed by the Global Assessment of Improvement Scale (GAI) modified form | 1 year
  The Global Assessment of Improvement Scale (GAI) modified form will assess Behcet disease's improvement of symptoms using a 7-point scale, with higher scores meaning an improvement of the symptoms. The severity of abdominal pain, severity of abdominal distention, satisfaction with bowel habits, severity of headache, severity of exhaustion, severity of nausea, attention disorder, muscle/joint pain, and quality of life will be investigated in response to the following question: "Compared to the way you felt before you entered the study, have your symptoms over the past 7 days been: 1) "Substantially Worse", 2) "Moderately Worse, 3) "Slightly Worse", 4) "No Change", 5) "Slightly Improved", 6) "Moderately Improved" or 7) "Substantially Improved".
Behcet disease's severity of gastrointestinal symptoms assessed by the Symptom Severity Scale (SSS) modified form | 1 year
  The Symptom Severity Scale (SSS) modified form is a multidimensional rating scale assessing overall symptoms' severity on a Visual Analogue Scale (VAS). An overall score will be calculated from six items: pain severity, pain frequency, abdominal bloating, bowel habit dissatisfaction, abdominal heaviness, and life interference. The modified SSS ranges from 0 to 600, with higher scores meaning more severe symptoms.

SECONDARY OUTCOMES:
Gut microbiota assessed by Illumina MiSeq platform | 1 year
  Changes of gut microbiota profiles from baseline. The V3 and V4 hypervariable regions of the 16S rRNA gene will be sequenced on Illumina MiSeq platform, following the Illumina protocol for 16S Metagenomic Sequencing Library Preparation
Fecal SCFA assessed by Gas Chromatography - Mass Spectrometry system | 1 year
  Fecal SCFA's change from baseline, especially butyrate, will be assessed by Gas Chromatography - Mass Spectrometry system
Inflammatory profile assessed by cytofluorimetric approach | 1 year
  Inflammatory cytokines' change from baseline, will be assessed with the Bio-Plex cytokine assay, according to the manufacturer's instructions. In particular, Interleukin (IL)-1ra (pg/mL), IL-4 (pg/mL), IL-6 (pg/mL), IL-8 (pg/mL), IL-10 (pg/mL), IL-12 (pg/mL), IL-17 (pg/mL), monocyte chemoattractant protein (MCP)-1 (pg/mL), macrophage inflammatory protein (MIP)-1beta (pg/mL), vascular endothelial growth factor (VEGF) (pg/mL), tumor necrosis factor (TNF)-alpha (pg/mL), interferon (IFN)-gamma (pg/mL), interferon-gamma-induced protein (IP)-10 (pg/mL), will be measured.
Lipid peroxidation assessed by flow cytometry | 1 year
  Lipid peroxidation markers' change from baseline will be estimated using the Thiobarbituric Acid Reactive Substances (TBARS, pg/mL) assay kit through the flow cytometry.
Plasma total antioxidant capacity assessed by the oxygen radical absorbance capacity | 1 year
  Plasma total antioxidant capacity's (TAC, μmol/mL) change from baseline, will be measured using the oxygen radical absorbance capacity.
Reactive oxygen species (ROS) assessed by flow cytometry | 1 year
  Leukocyte (lymphocyte, monocyte, and granulocyte) reactive oxygen species' (ROS, RFU) change from baseline will be assessed through flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Casini, MD, Study Director — Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy
Locations (1):
- Unit of Clinical Nutrition, University Hospital of Careggi, Florence, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Skef W, Hamilton MJ, Arayssi T. Gastrointestinal Behcet's disease: a review. World J Gastroenterol. 2015 Apr 7;21(13):3801-12. doi: 10.3748/wjg.v21.i13.3801. PMID 25852265
- [Background] Consolandi C, Turroni S, Emmi G, Severgnini M, Fiori J, Peano C, Biagi E, Grassi A, Rampelli S, Silvestri E, Centanni M, Cianchi F, Gotti R, Emmi L, Brigidi P, Bizzaro N, De Bellis G, Prisco D, Candela M, D'Elios MM. Behcet's syndrome patients exhibit specific microbiome signature. Autoimmun Rev. 2015 Apr;14(4):269-76. doi: 10.1016/j.autrev.2014.11.009. Epub 2014 Nov 27. PMID 25435420
- [Background] Neish AS. Microbes in gastrointestinal health and disease. Gastroenterology. 2009 Jan;136(1):65-80. doi: 10.1053/j.gastro.2008.10.080. Epub 2008 Nov 19. PMID 19026645
- [Background] Candela M, Rampelli S, Turroni S, Severgnini M, Consolandi C, De Bellis G, Masetti R, Ricci G, Pession A, Brigidi P. Unbalance of intestinal microbiota in atopic children. BMC Microbiol. 2012 Jun 6;12:95. doi: 10.1186/1471-2180-12-95. PMID 22672413
- [Background] Kosiewicz MM, Dryden GW, Chhabra A, Alard P. Relationship between gut microbiota and development of T cell associated disease. FEBS Lett. 2014 Nov 17;588(22):4195-206. doi: 10.1016/j.febslet.2014.03.019. Epub 2014 Mar 26. PMID 24681103
- [Background] Wong JM. Gut microbiota and cardiometabolic outcomes: influence of dietary patterns and their associated components. Am J Clin Nutr. 2014 Jul;100 Suppl 1:369S-77S. doi: 10.3945/ajcn.113.071639. Epub 2014 Jun 4. PMID 24898225
- [Background] Sonnenburg ED, Sonnenburg JL. Starving our microbial self: the deleterious consequences of a diet deficient in microbiota-accessible carbohydrates. Cell Metab. 2014 Nov 4;20(5):779-786. doi: 10.1016/j.cmet.2014.07.003. Epub 2014 Aug 21. PMID 25156449
- [Background] Kabeerdoss J, Devi RS, Mary RR, Ramakrishna BS. Faecal microbiota composition in vegetarians: comparison with omnivores in a cohort of young women in southern India. Br J Nutr. 2012 Sep 28;108(6):953-7. doi: 10.1017/S0007114511006362. Epub 2011 Dec 20. PMID 22182464
- [Background] Haro C, Montes-Borrego M, Rangel-Zuniga OA, Alcala-Diaz JF, Gomez-Delgado F, Perez-Martinez P, Delgado-Lista J, Quintana-Navarro GM, Tinahones FJ, Landa BB, Lopez-Miranda J, Camargo A, Perez-Jimenez F. Two Healthy Diets Modulate Gut Microbial Community Improving Insulin Sensitivity in a Human Obese Population. J Clin Endocrinol Metab. 2016 Jan;101(1):233-42. doi: 10.1210/jc.2015-3351. Epub 2015 Oct 27. PMID 26505825
- [Background] Candela M, Biagi E, Soverini M, Consolandi C, Quercia S, Severgnini M, Peano C, Turroni S, Rampelli S, Pozzilli P, Pianesi M, Fallucca F, Brigidi P. Modulation of gut microbiota dysbioses in type 2 diabetic patients by macrobiotic Ma-Pi 2 diet. Br J Nutr. 2016 Jul;116(1):80-93. doi: 10.1017/S0007114516001045. Epub 2016 May 6. PMID 27151248
- [Background] Candela M, Maccaferri S, Turroni S, Carnevali P, Brigidi P. Functional intestinal microbiome, new frontiers in prebiotic design. Int J Food Microbiol. 2010 Jun 15;140(2-3):93-101. doi: 10.1016/j.ijfoodmicro.2010.04.017. Epub 2010 Apr 24. PMID 20471127
- [Background] International Team for the Revision of the International Criteria for Behcet's Disease (ITR-ICBD). The International Criteria for Behcet's Disease (ICBD): a collaborative study of 27 countries on the sensitivity and specificity of the new criteria. J Eur Acad Dermatol Venereol. 2014 Mar;28(3):338-47. doi: 10.1111/jdv.12107. Epub 2013 Feb 26. PMID 23441863
- [Background] Munoz-Gonzalez I, Jimenez-Giron A, Martin-Alvarez PJ, Bartolome B, Moreno-Arribas MV. Profiling of microbial-derived phenolic metabolites in human feces after moderate red wine intake. J Agric Food Chem. 2013 Oct 2;61(39):9470-9. doi: 10.1021/jf4025135. Epub 2013 Sep 19. PMID 24010549
- [Derived] Pagliai G, Dinu M, Fiorillo C, Becatti M, Turroni S, Emmi G, Sofi F. Modulation of gut microbiota through nutritional interventions in Behcet's syndrome patients (the MAMBA study): study protocol for a randomized controlled trial. Trials. 2020 Jun 9;21(1):511. doi: 10.1186/s13063-020-04444-6. PMID 32517729